CLINICAL TRIAL: NCT05199233
Title: The Benefit of Mindfulness-Based Intervention Using A Wearable Wellness Brain Sensing Device (Muse-S™) in the Treatment of Post-Covid Symptoms
Brief Title: Mindfulness Intervention for Post-Covid Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ivana T Croghan, PhD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-009820
Record Dates: First submitted 2022-01-18; First posted 2022-01-20 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Post Acute Sequelae of SARS-CoV-2
Keywords: Covid-19; PASC; Pandemic; Meditation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: All subjects will receive and use the Muse S™ Headband system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Muse S™ Headband system for post-Covid Syndrome (Experimental): Subjects will utilize the Muse S™ Headband system at least 4 times per week for a minimum of 10 minutes each time over a period of 3 months (12 weeks).
  Interventions: Device: Muse S™ Headband system

INTERVENTIONS:
Device: Muse S™ Headband system — Clinical grade, headband style, wireless EEG (electroencephalogram is a test used to evaluate the electrical activity in the brain) system and designed to interact with a mobile device (smartphone or tablet).

SUMMARY:
The purpose of this study is to assess the feasibility of using a wearable brain-sensing wellness device (Muse-S) to potentially reduce stress and anxiety during Post-Covid, which is characterized by increased stress and anxiety.

DETAILED DESCRIPTION:
This study will answer the following questions: 1) will patients experiencing Long-Covid Syndrome utilize a wearable brain-sensing wellness device to potentially reduce stress and anxiety 2) does using this wearable brain-sensing wellness device help decrease stress and anxiety in patients who are experiencing Long-Covid Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Identified with one of 3 Post-Covid Syndrome (PASC) phenotypes at Mayo Clinic Rochester.
* Not pregnant by subject self-report at time of consent.
* Have the ability to provide informed consent.
* Have the ability to complete all aspects of this trial.
* Have access to an iPhone, iPad, or Android device.
* Have no contraindicating comorbid health condition which would interfere with the proper use of the Muse-SÔ system, as determined by the clinical investigators.

Exclusion Criteria:

* Used an investigational drug within the past 30 days.
* Anyone that is not on a stable dose of medication for anxiety, depression or sleep.
* Currently (within the past 3 weeks) been practicing mindfulness training on a weekly/regular basis.
* Currently (within 3 weeks) has been enrolled in another clinical or research program which intervenes on the patients' QOL, or stress.
* An unstable medical or mental health condition as determined by the physician investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Croghan, PhD, Principal Investigator — Mayo Clinic; Ryan Hurt, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Hurt RT, Ganesh R, Schroeder DR, Hanson JL, Fokken SC, Overgaard JD, Bauer BA, Thilagar BP, Aakre CA, Pruthi S, Croghan IT. Using a Wearable Brain Activity Sensing Device in the Treatment of Long COVID Symptoms in an Open-Label Clinical Trial. J Prim Care Community Health. 2025 Jan-Dec;16:21501319251325639. doi: 10.1177/21501319251325639. Epub 2025 Mar 12. PMID 40071827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Post-Covid Syndrome were recruited from the Long Covid Clinic at the Mayo Clinic Rochester Site.
Period: Overall Study
Arm/Group | Muse S™ Headband System for Post-Covid Syndrome
Started | 45
Completed | 44
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Muse S™ Headband System for Post-Covid Syndrome
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race/ethnicity: White, Non-Hispanic | 43
  race/ethnicity: other | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Stress
Description: Stress is evaluated through the Perceived Stress Scale (PSS). This is a 10-item Likert scale that measures global life stress by assessing the degree to which experiences are appraised as uncontrollable or unpredictable. Scores can range from 0 to 40, with higher scores indicating greater perceived stress. The outcome measure is change in stress from baseline at 3 months (end of treatment). Negative changes indicate decreased stress relative to baseline.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Muse S™ Headband System for Post-Covid Syndrome
Number analyzed (Participants) | 45
units on a scale | -5.0 (5.3)
Statistical Analysis 1: Comparison: Muse S™ Headband System for Post-Covid Syndrome; Test type: Superiority; p < 0.001, t-test, 2 sided; The mean change from baseline was compared to zero using a one-sample t-test

2. Primary Outcome: Change in Anxiety
Description: PROMIS Emotional Distress-short form 7a (7 items). The PROMIS Anxiety item banks assess self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety. The raw scores were converted to t-scores using published guidelines (see PROMIS website). A T-score of 50 is the average for the general population with a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured; thus, an increase in emotional distress T score corresponds to more anxiety - which is a worse outcome.
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Muse S™ Headband System for Post-Covid Syndrome
Number analyzed (Participants) | 45
units on a scale | -4.5 (5.5)
Statistical Analysis 1: Comparison: Muse S™ Headband System for Post-Covid Syndrome; Test type: Superiority; p < 0.001, t-test, 2 sided; The mean change from baseline was compared to zero using a one-sample t-test

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Muse S™ Headband System for Post-Covid Syndrome
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 1/45
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Muse S™ Headband System for Post-Covid Syndrome (N=45)
migraine headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT05199233/Prot_SAP_000.pdf